CLINICAL TRIAL: NCT06521294
Title: Effect of the Mulligan SNAG Technique on Structure of Intervertebral Disc and Physical Functioning in Individuals With Lumbar Intervertebral Disc Protrusion: A Randomized Controlled Study
Brief Title: Mulligan SNAG Technique in Individuals With Lumbar Intervertebral Disc Protrusion
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Ugur Cavlak, CLINICAL PROFESSOR, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BiruniUniversity34
Record Dates: First submitted 2024-07-16; First posted 2024-07-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Intervertebral Disc Protrusion
Keywords: Lumbar disc herniation; Mulligan Snag technique; Low back pain; MRI; Physical Functioning; Quality of life
MeSH Terms: conditions — Intervertebral Disc Displacement; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): SNAG
  Interventions: Other: Mulligan SNAG mobilization tecnique; Other: Conventional Physiotherapy
- Group 2 (Active Comparator): Physiotherapy
  Interventions: Other: Conventional Physiotherapy

INTERVENTIONS:
Other: Mulligan SNAG mobilization tecnique — Mulligan SNAG mobilization tecnique
  Arms: Group 1
Other: Conventional Physiotherapy — Conventional Physiotherapy

SUMMARY:
This study aimed to examine the effects of the Mulligan SNAG mobilization technique, applied in addition to conventional physiotherapy on the structure of the intervertebral disc and physical functioning in patients diagnosed with low back pain due to lumbar intervertebral disc protrusion. 38 volunteer patients will participate in the study. The participants will be randomized as an interventional and control gropus.

DETAILED DESCRIPTION:
Participants will be treated 3 days a week for 4 weeks. The session duration will be 40-45 minutes. Visual analog scale-VAS, oswestry disability index, magnetic imaging-MRI assessment, functıonal independence scale-FIM, Tampa kinesiophobia scale, one leg stand test, sit-stand test, 10-meter walking test, cadence , Nottingham health profile will be used to assses the participants in the two groups. All participants will be evaluated in the 5th week of the study. The program includes physical therapy session (Hot packed, trans cuteneal electric stimulation, therapeutic ultrasound, and therapautic exercises) and the Mulligan SNAG mobilization technique.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 20-60
2. Those diagnosed with lumbar intervertebral disc heniation (protrusion on L1-L2, L2-L3, L3-L4, L4-L5, L5-S1) at a single level
3. Those who voluntarily agreed to participate in the study

Exclusion Criteria:

* Individuals diagnosed with Lumbar Bulging, Extruded, Sequestered discs
* Individuals who have undergone lumbar region spinal surgery
* Individuals with spinal deformity (scoliosis, spondylolisthesis, Ankylosing Spondylitis)
* Individuals with lumbar stenosis
* Pregnant women
* Individuals receiving treatment for malignancy (primary or metastatic tumoral conditions in the lumbar region)
* Individuals diagnosed with advanced osteoporosis
* Individuals diagnosed with discitis

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-02-16 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging | baseline and iafter the intervention (in the 5th week)
  to measure protrusion (bigger amount means worse outcome)
Visual Analog Scale-VAS | baseline and immediately after the intervention (in the 5th week)
  to measure pain intensity (min. score is 0 and max. score is 10- higher score means worse outcome)

SECONDARY OUTCOMES:
Oswestry Disability Index-ODI | baseline and immediately after the intervention (in the 5th week)
  to describe disabilty level resulting from pain (min. score is 0 and max. score is 50- higher score means worse outcome)
Functional Independence Measure- FIM | baseline and immediately after the intervention (in the 5th week)
  to measure independency in daily living activities (min. score is 18 and max score is 156- higger score means better independency in daily living activities)
Tampa Kinesiophobia Scale- TKS | baseline and immediately after the intervention (in the 5th week)
  to measure anxiety-avoidance state (min. score is 17 and max. score is 68- higher score means worse outcome)
One Leg stand Test- OLST | before and after the intervention (in the 5th week)
  to measure static balance ability (min. score 0 and max. score is 60- Higher score means better balance)
Sit-Stand Test-SST | before and after the intervention (in the 5th week)
  to measure lower extremity performance (min. score is 0 and max. score is 30- higher score means better outcome)
10-m Walking test and cadance measurement | before and after the intervention (in the 5th week)
  to measure walking speed (in second- higher score means worse outcome) and cadance (number of steps during the test- higher score means better outcome)
Nottingham Health profile-NHP | before and after the intervention (in the 5th week)
  to describe level of quality of life (min. score is 38 and max. score is 3800 - higher score means poor health)

CONTACTS AND LOCATIONS:
Overall Officials: UGUR CAVLAK, Prof., Principal Investigator — Biruni University
Locations (1):
- Faculty of Health Sciences in Biruni University, Istanbul, ZEYTINBURNU, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hussien HM, Abdel-Raoof NA, Kattabei OM, Ahmed HH. Effect of Mulligan Concept Lumbar SNAG on Chronic Nonspecific Low Back Pain. J Chiropr Med. 2017 Jun;16(2):94-102. doi: 10.1016/j.jcm.2017.01.003. Epub 2017 Mar 30. PMID 28559749